CLINICAL TRIAL: NCT07332286
Title: Mini-percutaneous Nephrolithotomy With a Flexible Mini-nephroscope and a Flexible and Navigable Suction Access Sheath for Complex Renal Stones: A Prospective Pilot Study
Brief Title: FANS-Assisted Mini-PCNL for Complex Renal Stones
Acronym: FANS-perc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice chairman, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-252-02; ES-2025-252-02 (Other: The First Affiliated Hospital of Guangzhou Medical University)
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones
Keywords: PCNL; FANS; kidney stone; mini-PCNL
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FANS-assisted mini-PCNL (Experimental): Mini-percutaneous nephrolithotomy performed using a flexible mini-nephroscope combined with a flexible and navigable suction access sheath to facilitate flexible access and active stone fragment evacuation.
  Interventions: Procedure: FANS-assisted mini-percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: FANS-assisted mini-percutaneous nephrolithotomy — The procedure consists of mini-percutaneous nephrolithotomy (mini-PCNL) performed with the assistance of a flexible mini-nephroscope and a flexible and navigable suction access sheath (FANS).
  Following standard percutaneous renal access and initial stone fragmentation using a rigid nephroscope, a flexible mini-nephroscope is introduced through the percutaneous tract to access calyces that are difficult to reach with rigid instruments. Holmium:YAG laser lithotripsy is then performed under flexible endoscopic visualization.
  The flexible and navigable suction access sheath allows simultaneous irrigation and adjustable negative-pressure suction, enabling continuous evacuation of stone fragments during lithotripsy. Suction strength can be regulated intraoperatively to maintain a clear endoscopic field and facilitate controlled fragment removal.
  This procedure is applied to all participants in this prospective pilot study and aims to evaluate the feasibility and safety of flexible suction
  Other Names: Mini-PCNL using a flexible mini-nephroscope with suction access sheath

SUMMARY:
This prospective pilot study aims to evaluate the feasibility, safety, and preliminary clinical outcomes of a novel mini-percutaneous nephrolithotomy (mini-PCNL) technique integrating a flexible mini-nephroscope with a flexible and navigable suction access sheath (FANS) for the treatment of complex renal stones.

Thirty consecutive patients with renal stones ≥2 cm will be prospectively enrolled. All patients will undergo FANS-assisted mini-PCNL. The primary outcome is the immediate stone-free rate assessed by non-contrast CT within 72 hours after surgery. Secondary outcomes include operative parameters, postoperative pain, complications, length of hospital stay, and quality of life.

This pilot study is designed to provide preliminary evidence supporting the feasibility and safety of FANS-assisted mini-PCNL and to inform the design of future larger-scale studies.

DETAILED DESCRIPTION:
Conventional mini-PCNL may be limited by restricted access to anatomically challenging calyces and inefficient evacuation of stone fragments when flexible nephroscopy is required.

A novel technique integrating a flexible mini-nephroscope with a flexible and navigable suction access sheath (FANS) has been developed to enable flexible intrarenal navigation combined with active suction during antegrade lithotripsy.

This prospective pilot study will enroll 30 consecutive patients undergoing FANS-assisted mini-PCNL for complex renal stones. The study focuses on feasibility, safety, and preliminary clinical outcomes, including stone clearance and perioperative morbidity. The results will serve as preliminary data for future confirmatory or comparative clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Patients with renal stones measuring 2 cm or larger in maximum diameter
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Planned to undergo mini-percutaneous nephrolithotomy
* Able and willing to provide written informed consent

Exclusion Criteria:

* Uncontrolled urinary tract infection at the time of surgery
* Known bleeding tendency or coagulation disorders
* Contraindication to general anesthesia
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Immediate stone-free rate | Postoperative day 0 to 3
  Absence of residual stones or fragments >2 mm detected by non-contrast CT

SECONDARY OUTCOMES:
Stone-free rate at 1 month | Postoperative day 30 (±7 days)
  Absence of residual stones or fragments >2 mm detected by non-contrast CT
Operative time | From skin puncture to completion of the procedure (intraoperative period)
  Total duration of the surgical procedure measured from puncture to completion of the operation
Postoperative pain score | Postoperative day 1
  Postoperative pain assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable.
Postoperative complications | Postoperative day 0 to 30
  Incidence and severity of postoperative complications classified according to the Clavien-Dindo grading system
Length of postoperative hospital stay | Postoperative day 0 to postoperative day 14
  Duration of hospital stay measured from completion of the procedure to hospital discharge
Quality of life score | Baseline and postoperative day 30
  Health-related quality of life assessed using the Wisconsin Stone Quality of Life (WISQOL) questionnaire, which consists of 28 items scored on a 5-point Likert scale. Total scores range from 0 to 140, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as this is a single-center prospective pilot study with a small sample size, and the data will be used primarily for exploratory and hypothesis-generating purposes.